CLINICAL TRIAL: NCT01431781
Title: A Prospective, Multi-center, Investigator Sponsored, Randomized Controlled Trial-- The Prophylactic Effect of Stilamin on Post-ERCP Pancreatitis
Brief Title: The Prophylactic Effect of Stilamin on Post-Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Digestive System Department in Changhai Hospital, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02324789755
Record Dates: First submitted 2011-09-07; First posted 2011-09-12 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Post-ERCP Acute Pancreatitis
MeSH Terms: interventions — Anti-Inflammatory Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stilamin+common daily treatment (Experimental)
  Interventions: Drug: Stilamin+common daily treatment
- common daily treatment (Active Comparator)
  Interventions: Other: Common daily practice

INTERVENTIONS:
Drug: Stilamin+common daily treatment — dose:250 micrograms bolus intravenous in 3 minutes when ERCP starts and continuous infusion for 11 hours after ERCP.
  Common daily treatment: fasted for 6h after ERCP, Fluid replacement, Gastric acid inhibition, Antiinflammatory.
  Other Names: Somatostatin:Stilamin
  Arms: stilamin+common daily treatment
Other: Common daily practice — Fasted for 6h after ERCP, Fluid replacement, Gastric acid inhibition, Antiinflammatory
  Other Names: Common daily practice including:; Fasted for 6h after ERCP,; Fluid replacement,; Gastric acid inhibition,; Antiinflammatory
  Arms: common daily treatment

SUMMARY:
Pancreatitis are one of the most common complications of post-ERCP (Endoscopic Retrograde Cholangiopancreatography), the incidence rate is 5&-10%, how to prevent PEP and hyperamylasemia is an important issue, somatostatin is widely used in the field of pancreas treatment. In order to explore the effects of somatostatin on prevent PEP(post-ERCP Pancreatitis), 908 subjects will be enrolled in two group in the study, one group is given common treatment, the other uses somatostatin in the base of common treatment.

DETAILED DESCRIPTION:
A prospective, multi-center, investigator sponsored, randomized controlled trial, 15 sites join in in China, 908 subjects will be enrolled.

A descriptive analysis will be performed on primary endpoint, containing frequency of number and percentage of patients. A two proportion equality test will be conducted to explore whether incidence rates are different.

Descriptive statistics including number (N), mean, median, standard deviation, minimum and maximum, will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age > 18 years.
* Normal amylase level before undergoing ERCP.
* Signed inform consent form and agreed to follow-up on time.

Exclusion Criteria:

* Pregnancy or history of allergy to somatostatin.
* Renal insufficiency (Scr>177umol/L).
* Acute myocardial infarction within 3 months of the procedure.
* History of subtotal gastrectomy (Billroth II Method).
* Symptom of shock before undergoing ERCP, such as hypotension (systolic blood pressure < 90mmHg) or tachycardia (HR > 120 bpm).
* Medical or psychological condition that would not permit the patient to complete the study or sign the informed consent .
* Patients involved in other study within 60 days.
* Patients unfitted for the study by investigators.
* All contraindications to Stilamin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 908 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
the prophylaxis effect of Stilamin on post-ERCP pancreatitis | the incidence rate of PEP at 24 h after ERCP in two groups
  If the serum amylase of patients elevation and 3 times higher than the normal values after ERCP 24 hours, patients also have clinical symptoms, without other acute abdominal diseases,such as gastrointestinal perforation,acute cholecystitia and acute cholangitis and etc. In this condition, it will be defined PEP(post-ERCP pancreatitis).
  A descriptive analysis will be performed on primary endpoint, containing frequecency of number and percentage of patients. A two proportion equality test will be conducted to explore whether incidence rates are different.

SECONDARY OUTCOMES:
the prophylaxis effect of Stilamin in sub-groups of patient with high risk | PEP occurence rate at 24 h after ERCP at high-risk patients in two groups
  If the serum amylase of patients elevation and 3 times higher than the normal values after ERCP 24 hours in high risk patients, who also have clinical symptoms, without other acute abdominal diseases,such as gastrointestinal perforation,acute cholecystitia and acute cholangitis and etc. In this condition, it will be defined PEP(post-ERCP pancreatitis).
  Descriptive statistics will be produced for all continuous variables.Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.
compare Stilamin treated group with the other group on the incidence of hyperamylasemia/adverse events. | the incidence of hyperamylasemia/adverse events at 24 h after ERCP in two groups
  Hyperamylasemia will be defined as the serum amylase 3 times more than the upper normal values, without clinical symptoms.During the study, any unexpected medical issue will be called adverse event.
  Descriptive statistics will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Zh Li, Pro., Principal Investigator — Changhai Hospital; Jian Xi Wan, Pro., Principal Investigator — Shanghai First People Hospital; Bing Hu, Pro., Principal Investigator — Eastern Hepatobiliary Surgery Hospital; Feng Xi Zhang, Pro., Principal Investigator — Hangzhou First People Hospital; Ping Xi Zhou, Pro., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Tang Sh Han, Pro., Principal Investigator — Jiangsu Province of TCM; Xun Ren, Pro., Principal Investigator — The People' Hospital of Heilongjiang Province; Gang Xu Guo, Pro., Principal Investigator — Xijing Hospital; Ping Bie, Pro., Principal Investigator — xinan hospital; An Di Tian, Pro., Principal Investigator — Tongji Hospital; Guo Zh Nie, Pro., Principal Investigator — Wulumuqi General Hospital of Chinese PLA; Ming Yi, Pro., Principal Investigator — Beijing Friendship Hospital; Hua Lo Lu, Pro., Principal Investigator — The First Affiliated Hospital of Nanchang University; Chao Fa Zhi, Pro., Principal Investigator — Nanfang Hospital, Southern Medical University; Ping Li He, Pro., Principal Investigator — Fujian Province Hospital
Locations (15):
- China (15):
  - Fujian Province Hospital, Fuzhou, Fujian
  - Nanfang Hospital, Guangzhou, Guangdong
  - The People' Hospital of Heilongjiang Province, Haerbin, Heilongjiang
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Xijing Hospital, Xi’an, Shanxi
  - Wulumuqi General Hospital of Chinese PLA, Ürümqi, Xinjiang
  - Hangzhou First People Hospital, Hangzhou, Zhejiang
  - Beijing Friendship Hospital, Beijing
  - Xinan Hospital, Chongqing
  - Jiangsu Province of TCM, Nanjing
  - Changhai Hospital, Shanghai
  - Eastern Hepatobiliary Surgery Hospital, Shanghai
  - Shanghai First People Hospital, Shanghai
  - Tongji Hospital, Wuhan

REFERENCES:
- [Derived] Bai Y, Ren X, Zhang XF, Lv NH, Guo XG, Wan XJ, Nie ZG, Han ST, Bie P, Tian DA, Ji M, Li ZS. Prophylactic somatostatin can reduce incidence of post-ERCP pancreatitis: multicenter randomized controlled trial. Endoscopy. 2015 May;47(5):415-20. doi: 10.1055/s-0034-1391227. Epub 2015 Jan 15. PMID 25590178